CLINICAL TRIAL: NCT06780267
Title: Clinical Study on Safety and Efficacy of HRS-2129 for Postoperative Analgesiain Orthopaedics
Brief Title: Clinical Study of HRS-2129 for Postoperative Analgesia in Orthopaedics
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-2129-103
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-01

CONDITIONS: Postoperative Pain in Orthopaedics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group: low\middle\high-dose (Experimental): HRS-2129； HRS-2129 placebo
  Interventions: Drug: HRS-2129; Drug: HRS-2129 placebo
- Treatment group:placebo (Experimental): HRS-2129 placebo
  Interventions: Drug: HRS-2129 placebo
- Treatment group: positive control (Active Comparator): Tramadol Hydrochloride SR Tablets
  Interventions: Drug: Tramadol Hydrochloride SR Tablets

INTERVENTIONS:
Drug: HRS-2129 — HRS-2129
  Arms: Treatment group: low\middle\high-dose
Drug: HRS-2129 placebo — HRS-2129 placebo
  Arms: Treatment group: low\middle\high-dose; Treatment group:placebo
Drug: Tramadol Hydrochloride SR Tablets — Tramadol Hydrochloride SR Tablets
  Arms: Treatment group: positive control

SUMMARY:
The study is being conducted to evaluate the safety, and efficacy of HRS-2129 for Postoperative analgesia in orthopaedics. To explore the reasonable dosage of HRS-2129 for Postoperative analgesia in orthopaedics.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Subjects requiring elective orthopedic surgery
3. Conform to the ASA Physical Status Classification

Exclusion Criteria:

1. Subjects with a history of severe allergies
2. Subjects with nervous system disease
3. Subjects with a history of mental illness
4. Subjects with abnormal liver and renal function
5. Subjects with poorly controlled hypertensive or hypotensive
6. QTc：>450ms（male），>470ms（female）
7. Subjects who screened positive for substance abuse
8. History of cardiac dysrhythmias requiring anti-arrhythmia treatment(s)
9. The investigators determined that other conditions were inappropriate for participation in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Safety：Incidence and severity of AE/SAE | from ICF signing date to day 12 since last dose(14 days)

SECONDARY OUTCOMES:
the Sum of Pain Intensity Differences in Pain Score Over 6hour、12hour、16hour、24hour、48hour、12hour-24hour、24hour-48hour under static and moving condition | 48hours
The response rate of NRS scores under static and moving condition at 24hour and 48hour after the first dose of medication | 48hours
Participant ' satisfaction score for analgesia treatment | 48hours
Investigator satisfaction score for analgesia treatment | 48hours
Time of first use of remedial analgesic medication | 48hours
Cumulative use of remedial analgesics | 48hours
Cmax | 5 days
Tmax | 5 days
AUC0-12h | 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Academy of Medical Sciences - Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided